CLINICAL TRIAL: NCT00352937
Title: Comparison of Cardiac Computed Tomography for the Detection of Coronary Artery Disease With Nuclear Stress Test
Status: Completed | Type: Observational
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Wen-Chih Wu, Staff Cardiologist, Providence VA Medical Center
Other Study IDs: 1124528
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary Arteriosclerosis; Tomography, X-Ray Computed; Tomography, Emission-Computed, Single-Photon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To compare the efficacy of 16-row multi-detector CT (MDCT) with standard myocardial perfusion imaging in detecting coronary artery disease (CAD) in patients without a previously established diagnosis of CAD.

DETAILED DESCRIPTION:
Nuclear stress testing is currently the established non-invasive modality in detecting flow-obstructing coronary artery disease (CAD).

Recently, multi-detector CT (MDCT) has emerged as a new modality that offers a non-invasive means to directly visualize coronary anatomy and any CAD. Studies have shown that MDCT has excellent sensitivity and a high negative predictive value in detecting significant CAD.

The purpose of this study is to compare MDCT with nuclear stress testing for detecting CAD in previously undiagnosed patients.

ELIGIBILITY:
Inclusion Criteria:

* Referred for a clinical indicated stress SPECT MPI
* Adequate IV access in both arms

Exclusion Criteria:

* History of coronary angioplasty or stent placement
* History of coronary bypass surgery
* Angiographic history of flow-limiting CAD
* Documented history of elevated cardiac markers
* Documented history of injury or infarct on ECG
* Absence of sinus rhythm
* Current history of renal insufficiency
* Known allergy to contrast dye
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients without prior CAD referred for nuclear stress testing
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Calcium score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih Wu, MD, Principal Investigator — Providence VAMC; Victor H Shin, MD, Principal Investigator — Providence VAMC
Locations (1):
- Providence Veterans Affairs Medical Center, Providence, Rhode Island, United States